CLINICAL TRIAL: NCT06665256
Title: A Phase 2, Randomized, Open-label, Controlled Study to Evaluate the Efficacy and Safety of Rapcabtagene Autoleucel Versus Comparator in Participants With Severe Refractory Idiopathic Inflammatory Myopathies (IIM)
Brief Title: Phase 2 Study of Rapcabtagene Autoleucel in Myositis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CYTB323L12201
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Idiopathic Inflammatory Myopathies
Keywords: Chimeric Antigen Receptor T cells (CAR-T); rapcabtagene autoleucel; idiopathic inflammatory myopathies (IIM); dermatomyositis; Anti-Synthetase Syndrome; Immune-Mediated Necrotizing Myopathy; Interstitial Lung Disease
MeSH Terms: conditions — Myositis; Dermatomyositis; Lung Diseases, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rapcabtagene autoleucel (Experimental): Single infusion of rapcabtagene autoleucel (YTB323)
  Interventions: Biological: Rapcabtagene autoleucel
- Comparator (Active Comparator): Investigator choice of treatment as per protocol
  Interventions: Other: Active Comparator Option

INTERVENTIONS:
Biological: Rapcabtagene autoleucel — Single infusion of rapcabtagene autoleucel after lymphodepleting therapy with fludarabine (adjusted based on renal impairment) and cyclophosphamide daily for 3 days.
  Other Names: YTB323
  Arms: Rapcabtagene autoleucel
Other: Active Comparator Option — Investigator choice of treatment as per protocol
  Arms: Comparator

SUMMARY:
A Phase 2, randomized, open-label, controlled study to evaluate the efficacy and safety of rapcabtagene autoleucel versus comparator in participants with severe refractory idiopathic inflammatory myopathies (IIM)

DETAILED DESCRIPTION:
This is a Phase 2, randomized, active-controlled study. This study comprises two cohorts:

* A lead-in cohort enrolling participants to receive rapcabtagene autoleucel
* A randomized cohort with participants receiving either rapcabtagene autoleucel or a comparator option.

Participants in the comparator arm whose signs and symptoms are not fully controlled may receive rapcabtagene autoleucel treatment once the participant is confirmed to be eligible

After end of study (EOS), participants who received rapcabtagene autoleucel infusion will enter a long-term follow-up (LTFU) period after rapcabtagene autoleucel infusion. This LTFU will be described in a separate study protocol.

ELIGIBILITY:
Key Inclusion Criteria:

1. Men and women, aged ≥ 18 and ≤75 years, with a diagnosis of probable or definite myositis according to American College of Rheumatology/European League Against Rheumatism 2017 (ACR/EULAR 2017) criteria
2. Participants who had inadequate response to prior therapy
3. Diagnosed with active disease
4. Participant must meet criteria for severe myositis

Key Exclusion Criteria:

1. Any condition during Screening that could prevent a complete washout of medications or could otherwise make the participant ineligible for anti-CD19 CAR-T therapy and further participation in the study
2. BMI at Screening of ≤17 or ≥40 kg/m2
3. Severe muscle damage at Screening
4. Inadequate organ function
5. Hypersensitivity and/or contraindications to any product (including its ingredients) to be given to the participant as per the study protocol
6. Other inflammatory and non-inflammatory myopathies
7. Any medical conditions that are not related to IIM that would jeopardize the ability of the participant to tolerate CD19 CAR-T cell therapy

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2029-07-17 (Estimated); Study Completion 2030-07-17 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving moderate- to-major improvement in Total Improvement Score (TIS) at Week 52 | Week 52
  The percentage of participants with a TIS of at least 40 at the 52nd week after the start of the study, corresponding to moderate-to-major improvement.

SECONDARY OUTCOMES:
Adjusted annual cumulative glucocorticoid dose up to Week 52 | Week 52
  The total amount of glucocorticoids administered over the course of a year measured up to the 52nd week of treatment.
Change from baseline in percent predicted Forced Vital Capacity (FVC%) at Week 52 | Baseline, Week 52
  The difference in the percentage of the predicted Forced Vital Capacity (FVC) from the start of the study to the 52nd week.
Proportion of participants achieving major improvement in TIS at Week 52 | Week 52
  The percentage of participants with a TIS of at least 60 at the 52nd week after the start of the study, corresponding to at least major improvement.
Change from baseline in Patient-Reported-Outcome Measurement Information System (PROMIS)-Fatigue 7a at Week 52 | Baseline, Week 52
  The difference in the fatigue levels reported by participants from the start of the study to the 52nd week.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (51):
- United States (5):
  - University Of Alabama, Birmingham, Alabama
  - FL Medical Clinic Orlando Health, Zephyrhills, Florida
  - Northwestern University, Chicago, Illinois
  - University Of Iowa, Iowa City, Iowa
  - LDS Hospital, Salt Lake City, Utah
- France (5):
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rennes
- Germany (8):
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Ulm
- Israel (3):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (3):
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Milan, MI
- Japan (10):
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Yokohama, Kanagawa-ku
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Izumo, Shimane
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Kyoto
- Novartis Investigative Site, Amsterdam, North Holland, Netherlands
- Novartis Investigative Site, Riyadh, Saudi Arabia
- Novartis Investigative Site, Singapore, Singapore
- Spain (8):
  - Novartis Investigative Site, Santiago Compostela, A Coruna
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Salamanca
- Novartis Investigative Site, Geneva, Switzerland
- Taiwan (3):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
- United Kingdom (2):
  - Novartis Investigative Site, Sheffield, South Yorkshire
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com